CLINICAL TRIAL: NCT07247773
Title: Turkish Validity and Reliability of CyberSickness in Virtual Reality Questionnaire
Brief Title: Turkish Adaptation of the CSQ-VR
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, enes tayyip benli, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-BENLI-008
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers
Keywords: Virtual Reality; Cybersickness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteer: A group of healthy participants will rate the symptoms induced in virtual reality using questionnaire items.

SUMMARY:
The Cybersickness in Virtual Reality Questionnaire (CSQ-VR) is a tool designed to measure the presence and intensity of cybersickness symptoms experienced in VR. The CSQ-VR is an adapted and improved version of the Cybersickness section of the Virtual Reality Neuroscience Questionnaire (VRNQ). The aim of this study is to examine the validity and reliability of the Turkish version of the CSQ-VR.

DETAILED DESCRIPTION:
Alongside the many innovations brought by virtual reality, some users may experience the phenomenon of cybersickness. Symptoms of cybersickness include nausea, disorientation, and oculomotor disturbances. Although cybersickness shares similarities with simulator sickness, it differs in terms of the frequency and severity of symptoms. In particular, users who experience cybersickness report increased overall discomfort due to nausea and disorientation. Cybersickness is also distinct from motion sickness, as cybersickness is triggered by visual stimulation, whereas motion sickness is induced by actual physical movement.

Although there is no comprehensive theoretical framework for cybersickness, the most common and dominant explanation is the sensory conflict theory. This framework suggests that the symptomatology of cybersickness arises from a sensory conflict between the vestibular (inner ear) and visual systems. Simply put, the perception of postural balance depends on a combination of visual, vestibular, and proprioceptive inputs. It is assumed that conflicting motion perception cues from these systems cause cybersickness. The technological source of this conflict is vection, an illusory sense of self-motion induced in VR. Vection is considered one of the main causes of cybersickness in VR. In particular, movements such as linear and angular accelerations are reported to provoke cybersickness in users.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to participate in the study
* Ability to stand and walk independently

Exclusion Criteria:

* Presence of amblyopia, strabismus, or pathologies impairing focus, depth perception, or normal 3D vision
* Failure on the butterfly test of the Titmus stereotest

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers aged 18-30 years with independent standing and walking ability will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Cybersickness in Virtual Reality Questionnaire | Immediately after a single VR session (~1 hour)
  It is a tool designed to measure the presence and severity of cybersickness symptoms experienced in VR

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire | Immediately after a single VR session (~1 hour)
  The Simulator Sickness Questionnaire evaluates 16 symptoms such as eye strain, nausea, sweating, and headache, each rated on four severity levels (none, slight, moderate, and severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, individual participant data (IPD) will not be made available to other researchers.